CLINICAL TRIAL: NCT02432261
Title: A Randomized, Two Center, Double-Blind Trial to Evaluate the Pharmacokinetics and Gonadotropin Suppression of Nestorone®-Testosterone (NES/T) Combination Gel in Healthy Men
Brief Title: Evaluate the Pharmacokinetics and Gonadotropin Suppression of Nestorone®-Testosterone (NES/T) Combination Gel in Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kimberly Myer (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Kimberly Myer, Program Director, Premier Research
Organization: Premier Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CCN005A
Record Dates: First submitted 2015-03-19; First posted 2015-05-04 (Estimated); Results first posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: spermatogenesis; androgen; male contraception
MeSH Terms: interventions — ST 1435; Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): 5.0 mL of the 1.62% Nestorone® /testosterone gel (containing 8.3 mg NES + 62.5 mg T) applied each day on the arms and shoulders
  Interventions: Drug: Nestorone® /testosterone gel
- Group 2 (Experimental): 4.4 mL of the 1.62% Testosterone only gel (AndrogelTM) (containing 62.7 mg T) applied each day to the arms and shoulders
  Interventions: Drug: Testosterone only gel

INTERVENTIONS:
Drug: Nestorone® /testosterone gel — Nestorone® /testosterone combined gel
  Arms: Group 1
Drug: Testosterone only gel — Testosterone only gel
  Other Names: Androgel
  Arms: Group 2

SUMMARY:
This is a prospective, randomized, double-blinded, two-center trial to evaluate the gonadotropin suppressive activity of transdermal treatment with a combined NES/T gel, or T gel alone, for 28 days.

DETAILED DESCRIPTION:
A total of 45 subjects will be enrolled and randomized in a 2:1 ratio to one of two treatment groups. A description of each group is as follows:

* Group 1 (30 subjects): 5.0 mL of the 1.62% combined gel (containing 8.3 mg NES + 62.5 mg T) applied each day on the arms and shoulders
* Group 2 (15 subjects): 4.4 mL of the 1.62% AndrogelTM (containing 62.7 mg T) applied each day to the arms and shoulders

The total duration of treatment will be 28 days followed by a 72 hour sampling period to assess half-life and a recovery period of at least 28 days, at which point the subjects will return to the clinic for an end of study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male volunteers in good health as confirmed by physical examination, medical history, and clinical laboratory tests of blood and urine at the time of screening;
2. 18 to 50 years of age;
3. BMI < 33 calculated as weight in Kg/(height in cm)2;
4. No history of hormonal therapy use in the last six months prior to the first screening visit;
5. Subject will agree to use a recognized effective method of contraception with his partner (i.e. at a minimum, condom for the male partner and an effective contraception for the female partner) during the course of the study treatment and recovery phase;
6. In the opinion of the investigator, subject is able to comply with the protocol, understand and sign an informed consent and HIPAA form;
7. Does not meet any of the exclusion criteria.
8. Sperm concentration ≥ 15 million sperm per milliliter ejaculate.

Exclusion Criteria:

1. Men participating in another clinical trial involving an investigational drug within the last 30 days prior to the first screening visit;
2. Men not living in the catchment's area of the clinic or within a reasonable distance from the site;
3. Clinically significant abnormal physical findings at screening;
4. Elevated PSA (levels ≥ 4 ng/mL), according to local laboratory normal values;
5. Abnormal serum chemistry values, according to local laboratory normal values that indicate liver or kidney dysfunction or that may be considered clinically significant;
6. Use of androgens or body building substances within 6 months before first screening visit;
7. Diastolic blood pressure (DBP) > 80 and/or Systolic (SBP) > 130 mm Hg;
8. EKG abnormal and clinically significant and QTC level longer than 450msec;
9. History of hypertension, including hypertension controlled with treatment;
10. Known history of primary testicular disease or disorders of the hypothalamic-pituitary axis;
11. Known hypersensitivity to progestins or androgen;
12. Family or personal history of venous thromboembolism;
13. Benign or malignant liver tumors; active liver disease;
14. Known history of reproductive dysfunction including vasectomy or infertility;
15. Known history of cardiovascular, renal, hepatic or prostatic disease;
16. A serious systemic disease such as diabetes mellitus or morbid obesity (body weight greater than 120% of ideal body weight or BMI limitation as above);
17. Known or suspected alcoholism or drug abuse that may affect metabolism/transformation of steroid hormones and study treatment compliance;
18. Known dermatitis or severe skin disorder;
19. Moderate or severe depression as determined by PHQ-9 score >15;
20. Partner is known to be pregnant;
21. Known or suspected breast or prostate cancer;
22. Allergic to any ingredient in testosterone/nestorone gel, including alcohol;
23. Known history of untreated sleep apnea;
24. International Prostate Symptom Score (IPSS) greater than or equal to 15.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Wang, MD, Principal Investigator — Research Site; William Bremner, MD, Principal Investigator — Research Site
Locations (2):
- United States (2):
  - LA Biomedical Research Institute, Torrance, California
  - University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 29 | 15
Completed | 28 | 12
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 29 | 15 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 15 | 44
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (9.32) | 30.7 (7.29) | 32.7 (8.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 29 | 15 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 2 | 11
  Not Hispanic or Latino | 20 | 12 | 32
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 6 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 16 | 6 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 29 | 15 | 44

OUTCOME MEASURES:

1. Primary Outcome: Gonadotropin Suppression
Description: To quantify the gonadotropin suppressive activity of 4 weeks daily therapy of a combination transdermal gel containing 8.3 mg Nestorone® (NES) gel and 62.5 mg (1.62%) testosterone (T) gel, and of T gel (1.62%) alone. Specifically, the proportion (and 95% CI) of men who suppress both gonadotropins (luteinizing hormone [LH] and follicle-stimulating hormone [FSH]) to ≤ 1 IU/L in each group, will be quantified.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 24 | 11
Participants | 16 | 1
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Superiority — We did not statistically power this study; p = 0.003, Fisher Exact; difference of proportion of subjects = 57.6 — The difference of proportion = NES/Testosterone - Testosterone

2. Secondary Outcome: Gonadotropin and Follicle-stimulating Hormone Suppression
Description: • To quantify the proportion (and 95% CI) of men who suppress both gonadotropins (luteinizing hormone [LH] and follicle-stimulating hormone [FSH]) to the detection limit of the assay in each group.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 24 | 11
Participants | 12 | 1

3. Secondary Outcome: Change in LH and FSH Concentrations
Description: • To quantify the median percent change from baseline to week 4 and interquartile range for serum gonadotropins (LH and FSH) concentrations for each treatment group.
Time Frame: 4 weeks
Measure: Median (Standard Deviation); unit: IU/L
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 24 | 11
IU/L
  LH | -94.55 (26.656) | -31 (37.638)
  FSH | -90.25 (24.349) | -23.1 (33.577)

4. Secondary Outcome: Acceptability and Satisfaction as Measured by the Contraceptive Gel Acceptability and Satisfaction Questionnaire by Comparing T and NES Serum Concentrations.
Description: A simple acceptability questionnaire used previously in male CCTN studies was administered at treatment Day 28 (28, 29) for subjects to answer questions about the acceptability of gel as a product and as a method for contraception over the preceding 4 weeks.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 28 | 13
Participants
  Overall satisfaction: Strongly disagree | 1 | 0
  Overall satisfaction: disagree | 1 | 0
  Overall satisfaction: undecided | 4 | 2
  Overall satisfaction: agree | 15 | 9
  Overall satisfaction: Strongly agree | 7 | 2

5. Secondary Outcome: T Serum Concentrations
Time Frame: 8 weeks
Population: The difference in numbers means there was missing data
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 29 | 15
ng/dL
  Testosterone Day 7 | 502.9 (409.20) | 674.9 (283.97)
  Testosterone Day 28: 0 minutes pre-dose: number analyzed (Participants) | 27 | 12
  Testosterone Day 28: 0 minutes pre-dose | 602.1 (476.57) | 828.1 (567.58)
  Testosterone Day 56 (recovery): number analyzed (Participants) | 29 | 13
  Testosterone Day 56 (recovery) | 594.47 (217.718) | 595.81 (205.938)

6. Secondary Outcome: Secondary Outcome # 6 Part 1a: A Composite Safety of the Combined Gel Determined by Outcomes of CBC (Hemoglobin)
Description: General composite safety as measured various times during the study by CBC-Hemoglobin
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 28 | 12
g/dl | 0.01 (0.924) | -0.18 (0.634)

7. Secondary Outcome: Assessing Sexual Function by Compare Gonadotropin Suppressive Activity of T and NES Against T Alone Through the Psychosexual Daily Questionnaire.
Description: Sexual activity was rated on a scale from 0 (not at all) to 7 (very high enjoyment/pleasure). Erections were rated on a scale of 0 (not satisfactory) to 7 (very satisfactory). Results are change from baseline to final treatment evaluation.
Time Frame: 4 weeks
Population: The difference in numbers means there was missing data in the questionnaire which caused some of the domains to have missing results while some domains could have a score calculated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 27 | 12
score on a scale
  Sexual Activity | -0.18 (1.483) | -0.17 (0.676)
  Erections: number analyzed (Participants) | 26 | 11
  Erections | -0.6 (2.47) | -0.1 (1.14)

8. Secondary Outcome: Secondary Outcome # 6 Part 2a: A Composite Safety of the Combined Gel Determined by Outcomes of Chemistry
Description: Change from baseline to final treatment evaluation-Total Cholesterol, Triglycerides, HDL
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 27 | 12
mg/dL
  Total Cholesterol | -5.8 (18.21) | -1.4 (19.10)
  Triglycerides | -12.2 (31.16) | -15.8 (26.14)
  HDL | -2.3 (7.65) | -1.8 (5.65)

9. Secondary Outcome: Secondary Outcome # 6 Part 3a: A Composite Safety of the Combined Gel Determined by Outcomes of Vitals (Blood Pressure)
Description: Change from baseline to final treatment evaluation
Time Frame: 4 weeks
Population: The difference in numbers means there was missing data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 28 | 14
mmHg
  Systolic BP | 2.8 (6.91) | -2.2 (8.08)
  Diastolic BP | 1.8 (6.57) | 0.1 (6.20)

10. Secondary Outcome: Secondary Outcome # 6 Part 4: A Composite Safety of the Combined Gel Determined by Outcomes of Physical Changes
Description: Change from baseline to final treatment evaluation
Time Frame: 4 weeks
Population: The difference in numbers means there was missing data.
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 28 | 13
participants
  Skin: Improved | 0 | 0
  Skin: No Change | 27 | 12
  Skin: Worsened | 1 | 1
  Heart: Improved | 0 | 0
  Heart: No Change | 28 | 13
  Heart: Worsened | 0 | 0
  Digital Rectal Exam: Improved: number analyzed (Participants) | 16 | 10
  Digital Rectal Exam: Improved | 0 | 0
  Digital Rectal Exam: No Change: number analyzed (Participants) | 16 | 10
  Digital Rectal Exam: No Change | 16 | 10
  Digital Rectal Exam: Worsened: number analyzed (Participants) | 16 | 10
  Digital Rectal Exam: Worsened | 0 | 0

11. Secondary Outcome: Secondary Outcome # 6 Part 5: A Composite Safety of the Combined Gel Determined by Outcomes of Psychosexual Questionnaires
Description: Change from baseline to final treatment evaluation. Sexual motivation was rated on a scale of 0 (none) to 7 (very high). Erections were rated on a scale of 0 (not satisfactory) to 7 (very satisfactory).
Time Frame: 4 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 27 | 12
units on a scale
  Sexual Motivation: Change from baseline to final treatment | 0.01 (1.765) | -0.24 (0.839)
  Erections: Change from baseline to final treatment: number analyzed (Participants) | 26 | 11
  Erections: Change from baseline to final treatment | -0.6 (2.47) | -0.1 (1.14)

12. Secondary Outcome: Secondary Outcome # 6 Part 3: A Composite Safety of the Combined Gel Determined by Outcomes of Patient Health Questionnaires
Description: PHQ-9 Total Score: Change from baseline to final treatment evaluation. The Patient Health Questionnaire (PHQ)-9 is a self-administered instrument for screening, monitoring and diagnosis of depression. This questionnaire can be used repeatedly to monitor improvement or worsening of symptoms. Scale range is from 0 (not at all) to 3 (nearly every day).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 28 | 13
score on a scale | 0.6 (1.73) | 0.7 (1.44)

13. Secondary Outcome: NES Serum Concentrations
Time Frame: 8 weeks
Population: The difference in numbers means there was missing data
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 29 | 15
pmol/L
  Nesterone Day 7 | 679.73 (716.884) | 9.26 (34.673)
  Nesterone Day 28: 0 minutes pre-dose: number analyzed (Participants) | 27 | 12
  Nesterone Day 28: 0 minutes pre-dose | 820.60 (706.619) | 20.70 (49.697)
  Nesterone Day 56 (recovery): number analyzed (Participants) | 29 | 13
  Nesterone Day 56 (recovery) | 13.03 (33.335) | 0 (0)

14. Secondary Outcome: Secondary Outcome # 6 Part 1b: A Composite Safety of the Combined Gel Determined by Outcomes of CBC (WBC)
Description: General composite safety as measured various times during the study by CBC - WBC
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: WBCs per microliter
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 28 | 12
WBCs per microliter | 0.182 (0.9772) | -0.548 (1.0023)

15. Secondary Outcome: Secondary Outcome # 6 Part 1c: A Composite Safety of the Combined Gel Determined by Outcomes of CBC (Hematocrit)
Description: General composite safety as measured various times during the study by CBC-Hematocrit
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percentage of blood
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 28 | 12
percentage of blood | 0.19 (2.650) | -0.58 (1.527)

16. Secondary Outcome: Secondary Outcome # 6 Part 2b: A Composite Safety of the Combined Gel Determined by Outcomes of Chemistry
Description: Change from baseline to final treatment evaluation-ALT, AST
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 27 | 12
IU/L
  ALT | -4.4 (7.89) | 0.1 (7.80)
  AST | -2.0 (9.59) | 1.6 (15.90)

17. Secondary Outcome: Secondary Outcome # 6 Part 3b: A Composite Safety of the Combined Gel Determined by Outcomes of Vitals (Weight)
Description: Change from baseline to final treatment evaluation
Time Frame: 4 weeks
Population: The difference in numbers means there was missing data.
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 28 | 12
lbs | 0.045 (3.8638) | 1.2 (3.6888)

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/15
Other Adverse Events (participants affected / at risk) | 10/29 | 5/15
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=29) | Group 2 (N=15)
DIARRHEA (General disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
APPLICATION SITE RASH (General disorders) | 1 (1) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0)
LOCALIZED INFECTION (Infections and infestations) | 1 (1) | 0 (0)
EXCORIATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periorbital contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SUNBURN (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
THERMAL BURN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
CONVULSION (Nervous system disorders) | 0 (0) | 1 (1)
HEADACE (Nervous system disorders) | 1 (1) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
LIBIDO DECREASED (Psychiatric disorders) | 0 (0) | 1 (1)
Varicocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No